CLINICAL TRIAL: NCT00908544
Title: NEW ERA STUDY - HIV and Eradication: A Multicenter, Open-label, Non-randomized Trial to Evaluate Treatment With Multi-drug Class (MDC) HAART and Its Impact on the Decay Rate of Latently Infected CD4+ T Cells Incl. Amendment 1.0
Brief Title: New Era Study: Treatment With Multi Drug Class (MDC) HAART in HIV Infected Patients
Acronym: NewEra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MUC Research GmbH (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); AbbVie (Industry); Pfizer (Industry); German Center for Infection Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUC_NewEra_3.3; 2008-002070-35 (EudraCT Number); 4034932 (Other: BfArM); 08101 (Other: Bayerische Landesärztekammer); ID 8879 (Other Grant/Funding Number: Pfizer); IISP #35576 (Other Grant/Funding Number: MSD)
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: HIV Infections
Keywords: HIV-infection; Primary HIV-infection; Proviral DNA; Eradication; Multi drug class HAART
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PHI-patients (Experimental): Patients with primary HIV infection (PHI) (see also "Eligibility") are immediately treated with 2 NRTI + 1 PI/r + Maraviroc + Raltegravir
  Interventions: Other: PHI-patients
- CHI-patients (Experimental): Patients with chronic HIV infection (CHI) and with suppressed plasma viral load for at least three years under continuous HAART (2 NRTI + 1 PI/r see also "Eligibility") intensified by Maraviroc + Raltegravir
  Interventions: Other: CHI-patients

INTERVENTIONS:
Other: PHI-patients — Treatment initiation with multi drug class (MDC) HAART. 2 NRTI + 1 PI/r + Maraviroc + Raltegravir
  Arms: PHI-patients
Other: CHI-patients — Treatment intensification of PI-based HAART with Maraviroc and Raltegravir. 2 NRTI + 1 PI/r + Maraviroc + Raltegravir
  Arms: CHI-patients

SUMMARY:
This is a multi-center, open-label, non-randomized proof-of-concept trial. Two cooperating HIV-specialized centres represented by Dr. med. Hans Jaeger and Prof. Dr. Johannes Bogner are planning to perform an IIT (investigator initiated trial) with the goal to eradicate HIV in N=40 HIV-infected patients with either primary infection or chronic infection and successful HAART (Highly Active Antiretroviral Treatment) of several years.

All patients will be started on a multi-drug HAART including two Nucleoside-Reverse-Transcriptase-Inhibitors (NRTI´s), one Protease-Inhibitor (PI), a CCR5-inhibitor and an Integrase-Inhibitor (INI). Decay of viral reservoirs like latently HIV-infected CD4+ T-cells will be monitored over time.

DETAILED DESCRIPTION:
1. Recruitment and Treatment:

Recruitment will be stratified according to stage of HIV-infection and pre-treatment:

* Stratum I (PHI patients):

Patients presenting with primary HIV infection

* Stratum II (CHR patients):

Chronically HIV-infected patients with suppressed plasma viral load for ≥36 months under continuous HAART (Highly Active Antiretroviral Therapy).

CHR and PHI patients will be treated with an antiretroviral combination of five approved substances (Multi-Drug Class HAART= MDC HAART). Every regimen will contain Maraviroc and Raltegravir.

MDC HAART consisting of:

2 NRTI + 1PI + 1 CCR5 antagonist (= Maraviroc; MVC) + 1 INI (= Raltegravir; RAL).

The patients of the PHI-group will be immediately treated with MDC HAART for a duration of ≥5-7 years.

The patients of the CHR-group will be treated with MDC HAART after a 6-month observational lead-in phase for measuring laboratory parameters. Then HAART will be intensified with the respective missing drug classes of MDC HAART (MVC+RAL). The respective treatment time will be 2 years up to a Maximum of 7 years from baseline.

Dosing of antiretrovirals including study drugs Raltegravir and Maraviroc will be according to standard dosing as outlined in respective product informations (attached).

* Patients will take Raltegravir 400 mg (one 400 mg tablet) PO b.i.d. (without regard to food). Raltegravir which can be taken at any time of day but should be taken at the same time each day.
* Patients will take Maraviroc 150 mg (one 150 mg tablet) PO b.i.d. (without regard to food) if the co-administered PI is RTV-boosted Lopinavir, RTV-boosted Atazanavir, RTV-boosted Saquinavir, RTV-boosted Darunavir. Patients will take Maraviroc 300 mg (two 150 mg tablets) PO b.i.d. (without regard to food ) if the co-administered PI is Fosamprenavir or Tipranavir

In both treatment groups NRTI´s or PI´s can be replaced by other NRTI´s or PI´s in case of intolerability or other reasons at the discretion of the investigator.

Other treatments which are initiated by the treating physicians and which may have a potential impact on viral reservoirs (like valproic acid) or immunomodulators will not be discouraged during the course of the study.

If new antiretroviral agents will be approved or available through expanded access programs during the course of the study that might be beneficial for a study patient at the discretion of the treating physician, the treatment regimen can be modified based on current knowledge (=addition of new antiretroviral agent or replacement of drugs of the regimen). Patients will not be excluded from the study unless they reach the virological endpoint.

2. Study Procedures:

Each potential patient has to be informed about the study contents by the investigator and to sign the informed consent if he/she wants to participate to the study.

Then Each patient will be assigned to a unique allocation number at the first screening visit. A single patient cannot be assigned to more than one allocation number. Allocation number will be provided by the coordinating study centre.

Patients who meet the eligibility requirements will start their medication at baseline.

Monitoring of patient safety will be performed at all study visits; Specific laboratory measures are performed at a single visit after month 6 in all patients.

Visit time schedule:

- PHI-group: Screening/Baseline, Month 1, Month 3, Month 6 and following half-yearly

- CHI-group: Month -6 (Screening), Month -3 (Pre-baseline), Baseline, Month 1, Month 6 and following half-yearly Post Tx visits after pre-mature and regular discontinuation (including HAART interruption due to eradication, as defined . Follow-up visits post Tx (PFU1, PFU2, PFU3) are foreseen at months 3, 6 and 12.

According to the New Era study protocol, treatment can be interrupted in case of reaching undetectability of HIV-1 RNA in plasma and proviral DNA in PMBC. Because there are needed more virologic, immunologic or genetic markers to better predict virus control after treatment interruption, an approved Amendment (MUC_NewEra_v3.3 Protocol: EudraCT: 2008-002070-35 date: 6.11.2014; approved (BfArM) on 04.02.2015) has foreseen to conduct one additional blood sampling with the aim to better characterize and discriminate the New Era patients in terms of immunologic, virologic and other laboratory parameters

3. Safety Management:

At all visits, safety measurements of clinical chemistry, hematology and virology and physical examination will be conducted. All adverse events will be recorded.

Treatment naïve (PHI) female patients of childbearing potential will have pregnancy test performed at Screening, Baseline, Month 1, Month 3, Month 6 and following half-yearly until Month 90.

Pretreated (CHI) female patients of childbearing potential will have pregnancy test performed at Screen, 6 Month prior to Baseline, 3 Month prior to Baseline, at Baseline, Month 1, Month 3, Month 6 and following half-yearly until Month 54.

Serious Adverse Events (SAE´s):

Any serious adverse experience, whether or not there is a suspected causal relationship to the investigational product (including death due to any cause), which occurs to any subject/patient entered into this study or within 14 days following cessation of treatment or within the established off therapy follow-up period for safety described in the protocol, whether or not related to the investigational product, must be reported within 24 hours to one of the individual(s) listed on the sponsor.

For all serious adverse experiences the Serious Adverse Experience/Pregnancy/Overdose Case Report Form (SAE Form) will be completed. In addition, every single SAE will be recorded at the respective study visit in the Case Report Form.

Each SAE will be fully investigated and, if drug related, a decision will be made as to whether the risk/benefit warrants the patient´s continuation in the study.

Suspected Unexpected Serious Adverse Reaction´s (SUSAR's):

The Sponsor will report all SUSARs according to the standards for reporting SUSARs which are defined in 'Detailed guidance on the collection, verification and presentation of adverse reaction reports arising from clinical trials on medicinal products for human use - April 2006' and in accordance with all applicable global laws and regulations. SUSAR reports will include all informations required according to the Council for International Organizations of Medical Sciences CIOMS I reporting form.

The Sponsor who is non-commercial and not Marketing Authorization Holder (MAH) for any of the Investigational Medicinal Products (IMPs) will report all relevant information about a suspected unexpected serious adverse reaction (SUSAR) which occurs during the course of a clinical trial and is fatal or life-threatening as soon as possible to competent authority (Bundesinstitut für Arzneimittel und Medizinprodukte, BfArM), the relevant Ethics Committees, the investigators and the manufacturers of the study drugs. This needs to be done not later than 7 days after the Sponsor was first aware of the reaction. Any additional relevant information should be sent within 8 days of the report.

A Sponsor will report unexpected serious adverse reaction (SUSAR) which is not fatal or life-threatening as soon as possible, and in any event not later that 15 days after the Sponsor is first aware of the reaction.

The sponsor will inform all investigators concerned of findings that could adversely affect the safety of study subjects. If appropriate, the information can be aggregated in a line listing of SUSARs in periods and the volume of SUSARs generated. This line listing should be accompanied by a concise summary of the evolving safety profile of the investigational medicinal product.

If a significant safety issue is identified, either upon receipt of an individual case report or upon review of aggregate data, the sponsor will issue as soon as possible a communication to all investigators.

A safety issue that impacts upon the course of the clinical study or development project, including suspension of the study program or safety-related amendments to study protocols should also be reported to the investigators.

Data Safety Monitoring Board (DSMB):

The study will be monitored by an independent external Data Safety Monitoring Board (DSMB)/ Data Monitoring Committee (DMB). The DSMB will provide recommendations to the Oversight Committee. The Oversight Committee (consisting of the sponsor and coordinating investigator Dr. med. Hans Jaeger and principal investigator Prof. Johannes Bogner) will provide the overall scientific direction for the trial, and will receive and decide on any recommendations made by the DSMB. The Oversight Committee must approve all scientific reports concerning the main findings of the trial. The membership, procedures, functions and responsibilities of the Oversight Committee and DSMB will be identified in the New Era DSMB Charter.

Annual Safety Report (ASR):

In addition to the expedited reporting required for SUSAR, Sponsor will submit once a year throughout the clinical trial (or on request) a safety report to the competent authority (BfArM), and the relevant Ethics Committees of the concerned Member States.

4. Data Analysis:

This proof-of-concept study using a small, targeted number of subjects is carried out to determine if eradication of HIV is possible. A design with a placebo was discouraged in the light of possible eradication. The chronically infected patients serve as their own controls. Prior to baseline, these patients are monitored while on persistently suppressive HAART lasting already for at least 36 months and then switched to multi-drug class HAART.

Based on the assumption, that MDC (multi-drug class) HAART with Raltegravir and Maraviroc leads to a mean reduction of at least one 1 log in patients with PHI and assuming a standard deviation of 1 and a 95% confidence interval (0.5-1.5 log) with a width of 1, the sample size is calculated at ≥16 (assumption of normal distribution).

Intensification of HAART with Raltegravir and Maraviroc in chronically infected HIV-patients may have similar effects (Ramratnam B, J Acquir Immune Defic Syndr 2004; 35:33-37). Sample size calculation can be used also for chronically infected HIV-patients.

A sample size of 40 patients (20 primary infected patients (Stratum I, PHI) and 20 chronically infected patients (Stratum II, CHR) was chosen. Drop-outs in the first 12 months will be replaced.

In the course of this study no gender specific differences are expected. The application of Maraviroc and Raltegravir does not differ in male and female patients. The proportion of male and female patients will probably be in accordance with the epidemiologic data in Germany.

Hypothesis:

The hypotheses of this study is, that with MDC HAART, a mean reduction in proviral DNA of 1 log can be achieved by 36 months.

Null hypotheses H0: Mean reduction of proviral DNA < 1 log. Alternative hypotheses H1: Mean reduction of proviral DNA ≥1 log Level of significance : 0.05 Statistical test: One-tailed paired t-test

The null hypotheses will be rejected if the p-value of the test is less than the significance level (0.05).

The null hypotheses will be accepted if the p-value of the test greater than 0.05.

Statistical Methods:

For accepting or rejecting the primary hypothesis (of the trial, one-tailed paired t-test will be used.

Performed analysis will be descriptive and explorative.

ELIGIBILITY:
1. Inclusion Criteria:

   For all patients:
   * HIV-infected patient
   * Age greater 18 years
   * No acute AIDS-defining disease or history of AIDS- defining disease
   * CD4-cell nadir above or equal 200 cells/µL
   * Hemoglobin greater 8 g/dl
   * Neutrophil count greater 750 cells/µL
   * Platelet count greater 50.000 cells/µL
   * AST/ALT below 5x upper limit of normal range
   * No evidence for drug intolerability
   * No prior use of an HIV integrase inhibitor or CCR5 antagonist
   * No presence of malignancy (requiring active treatment and malignancy within 5 years prior to enrolment (even if in complete remission)
   * No significant underlying disease (non-HIV) that might impinge upon disease progression or death
   * No history of alcohol or other substance abuse or other condition which in the opinion of the investigator would interfere with the patient compliance or safety.
   * Written informed consent
   * For males and premenopausal females use of acceptable methods of birth control during the entire study and for 6 weeks thereafter
   * No pregnancy (for premenopausal women: negative serum or urine pregnancy test within 48 hours prior to initiating study medications)
   * No breastfeeding

   For chronically HIV-infected patients (CHI):
   * Continuous plasma viral load below 50 copies/ml for the preceding 36 months under HAART (two or less single viral load blips up to 500 copies/ml are allowed)
   * Stable HAART (for at least 3 months) prior to the Screening visit consisting of 2 NRTI + 1 PI
   * No history of virological failure
   * No documented resistance to PI and NRTI
   * CCR5-tropic virus

   For patients with primary HIV infection (PHI):
   * Detectable plasma viral load
   * ELISA positive or negative and Western Blot negative or positive with less or equal 2 bands at screening visit
   * No primary resistance to PI´s and NRTI´s
   * CCR5-tropic virus
2. Exclusion criteria:

Evidence for drug intolerability or contraindication concerning any drug foreseen for MDC HAART

* Documented HIV-1 resistance to PI and/or NRTI.
* CD4 nadir <200/µL
* Acute AIDS-defining disease or history of AIDS-defining disease
* CHI: preceding virological failure
* History of alcohol or other substance abuse or other condition which in the opinion of the investigator would interfere with the patient compliance or safety.
* Any of the following abnormal laboratory test results in screening:

  1. Hemoglobin < 8 g/dL
  2. Neutrophil count < 750 cells/µL
  3. Platelet count < 50,000 cells/µL
  4. AST or ALT > 5x the upper limit of normal
* Presence of malignancy (requiring active treatment and malignancy within 5 years prior to enrolment (even if in complete remission)
* Significant underlying disease (non-HIV) that might impinge upon disease progression or death
* Prior use of any experimental HIV- Integrase-Inhibitor or CCR5-antagonist.
* Patient is pregnant or breastfeeding, or expecting to conceive (within the duration of the study). Patient is expecting to donate eggs (within the duration of the study). Patient is expecting to donate sperm (within the duration of the study).
* Contraindications for Maraviroc (Celsentri®) or Raltegravir (Isentress®) according to the respective summary of product characteristics (see also product informations attached to the protocol) (Hypersensitivity to the active substances or any of the excipients).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-05-15 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Jaeger, MD, Study Chair — MUC Research GmbH; Johannes Bogner, Prof., MD, Study Chair — University Munich, University Hospital, Dept. of Infectious Diseases,
Locations (8):
- Germany (8):
  - Onkology Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - Private Practice for Internal Medicine, Hematology and Oncology, Mannheim, Baden-Wurttemberg
  - Private Practice Drs Ulmer/Frietsch/Mueller, Stuttgart, Baden-Wurttemberg
  - Practice Dr. med. Lothar Schneider, Fürth, Bavaria
  - Private Practice Drs Pauli/Becker, Munich, Bavaria
  - MVZ Karlsplatz, Munich, Bavaria
  - University Munich University Hospital, Dept. of Infectious Diseases, Munich, Bavaria
  - ICH Study Center, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Mascio M, Dornadula G, Zhang H, Sullivan J, Xu Y, Kulkosky J, Pomerantz RJ, Perelson AS. In a subset of subjects on highly active antiretroviral therapy, human immunodeficiency virus type 1 RNA in plasma decays from 50 to <5 copies per milliliter, with a half-life of 6 months. J Virol. 2003 Feb;77(3):2271-5. doi: 10.1128/jvi.77.3.2271-2275.2003. PMID 12525664
- [Background] Lehrman G, Hogue IB, Palmer S, Jennings C, Spina CA, Wiegand A, Landay AL, Coombs RW, Richman DD, Mellors JW, Coffin JM, Bosch RJ, Margolis DM. Depletion of latent HIV-1 infection in vivo: a proof-of-concept study. Lancet. 2005 Aug 13-19;366(9485):549-55. doi: 10.1016/S0140-6736(05)67098-5. PMID 16099290
- [Background] Ramratnam B, Mittler JE, Zhang L, Boden D, Hurley A, Fang F, Macken CA, Perelson AS, Markowitz M, Ho DD. The decay of the latent reservoir of replication-competent HIV-1 is inversely correlated with the extent of residual viral replication during prolonged anti-retroviral therapy. Nat Med. 2000 Jan;6(1):82-5. doi: 10.1038/71577. PMID 10613829
- [Background] Sedaghat AR, Siliciano JD, Brennan TP, Wilke CO, Siliciano RF. Limits on replenishment of the resting CD4+ T cell reservoir for HIV in patients on HAART. PLoS Pathog. 2007 Aug 31;3(8):e122. doi: 10.1371/journal.ppat.0030122. PMID 17784786
- [Background] Sedaghat AR, Siliciano RF, Wilke CO. Low-level HIV-1 replication and the dynamics of the resting CD4+ T cell reservoir for HIV-1 in the setting of HAART. BMC Infect Dis. 2008 Jan 2;8:2. doi: 10.1186/1471-2334-8-2. PMID 18171475
- [Background] Siliciano JD, Kajdas J, Finzi D, Quinn TC, Chadwick K, Margolick JB, Kovacs C, Gange SJ, Siliciano RF. Long-term follow-up studies confirm the stability of the latent reservoir for HIV-1 in resting CD4+ T cells. Nat Med. 2003 Jun;9(6):727-8. doi: 10.1038/nm880. Epub 2003 May 18. PMID 12754504
- [Background] Zhang L, Ramratnam B, Tenner-Racz K, He Y, Vesanen M, Lewin S, Talal A, Racz P, Perelson AS, Korber BT, Markowitz M, Ho DD. Quantifying residual HIV-1 replication in patients receiving combination antiretroviral therapy. N Engl J Med. 1999 May 27;340(21):1605-13. doi: 10.1056/NEJM199905273402101. PMID 10341272
- [Background] Henrich TJ, Hanhauser E, Marty FM, Sirignano MN, Keating S, Lee TH, Robles YP, Davis BT, Li JZ, Heisey A, Hill AL, Busch MP, Armand P, Soiffer RJ, Altfeld M, Kuritzkes DR. Antiretroviral-free HIV-1 remission and viral rebound after allogeneic stem cell transplantation: report of 2 cases. Ann Intern Med. 2014 Sep 2;161(5):319-27. doi: 10.7326/M14-1027. PMID 25047577
- [Background] Hutter G, Ganepola S. Eradication of HIV by transplantation of CCR5-deficient hematopoietic stem cells. ScientificWorldJournal. 2011 May 5;11:1068-76. doi: 10.1100/tsw.2011.102. PMID 21552772
- [Background] Persaud D, Gay H, Ziemniak C, Chen YH, Piatak M Jr, Chun TW, Strain M, Richman D, Luzuriaga K. Absence of detectable HIV-1 viremia after treatment cessation in an infant. N Engl J Med. 2013 Nov 7;369(19):1828-35. doi: 10.1056/NEJMoa1302976. Epub 2013 Oct 23. PMID 24152233
- [Background] Saez-Cirion A, Bacchus C, Hocqueloux L, Avettand-Fenoel V, Girault I, Lecuroux C, Potard V, Versmisse P, Melard A, Prazuck T, Descours B, Guergnon J, Viard JP, Boufassa F, Lambotte O, Goujard C, Meyer L, Costagliola D, Venet A, Pancino G, Autran B, Rouzioux C; ANRS VISCONTI Study Group. Post-treatment HIV-1 controllers with a long-term virological remission after the interruption of early initiated antiretroviral therapy ANRS VISCONTI Study. PLoS Pathog. 2013 Mar;9(3):e1003211. doi: 10.1371/journal.ppat.1003211. Epub 2013 Mar 14. PMID 23516360
- [Result] Grutzner EM, Hoffmann T, Wolf E, Gersbacher E, Neizert A, Stirner R, Pauli R, Ulmer A, Brust J, Bogner JR, Jaeger H, Draenert R. Treatment Intensification in HIV-Infected Patients Is Associated With Reduced Frequencies of Regulatory T Cells. Front Immunol. 2018 Apr 30;9:811. doi: 10.3389/fimmu.2018.00811. eCollection 2018. PMID 29760693

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall 47 patients signed informed consent, of which 42 participated in the study; five patients turned out to be screening failures due to nonfulfillment of the eligibility criteria (tropism test showed X4 tropism in three patients or Western blot bands >2 in two patients).
Groups:
- CHI-patients: Patients with chronic HIV infection (CHI) and with suppressed plasma viral load for at least three years under continuous HAART (2 NRTI + 1 PI/r see also "Eligibility") intensified by Maraviroc + Raltegravir
  CHI-patients: Treatment intensification of PI-based HAART with Maraviroc and Raltegravir.
  2 NRTI + 1 PI/r + Maraviroc + Raltegravir
Period: Overall Study
Arm/Group | CHI-patients | PHI-patients
Started | 20 | 22
Completed | 15 | 16
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lack of Efficacy | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Relocation abroad | 1 | 1
Not completed — Unable to visit sutdy center | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety dataset (safety population) is based on all patients having received at least one dose of study drugs (N=47 pts.); 5 of these patients were excluded.
  The efficacy dataset (efficacy population) is based on patients who were enrolled in the study, received at least one dose of study drugs and met the inclusion criteria (N=42 pts.).
Groups:
- Total: Total of all reporting groups
Arm/Group | CHI-patients | PHI-patients | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43.3 [33.8 to 51.0] | 40.2 [29.4 to 42.7] | 41.0 [31.7 to 46.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 14 | 21 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 20 | 22 | 42
HIV DNA in PBMC (peripheral blood mononuclear cells) [Median (Inter-Quartile Range); unit: log copies/10^6 PBMC] — Population: One Patient of CHI-Group had no HIV DNA measurement.
  log copies/10^6 PBMC
    number analyzed (Participants) | 19 | 22 | 41
    (all) | 2.5 [0.2 to 2.7] | 3.6 [3.5 to 3.8] | 3 [2.5 to 3.6]
HIV DNA in CD4+T cells [Median (Inter-Quartile Range); unit: log copies/10^6 CD4+T cells] — Population: One Patient of CHI-Group had no HIV DNA measurement.
  log copies/10^6 CD4+T cells
    number analyzed (Participants) | 19 | 22 | 41
    (all) | 3 [2.6 to 3.3] | 4.4 [4.1 to 4.6] | 3.6 [3.1 to 4.4]
HIV RNA in Plasma [Median (Inter-Quartile Range); unit: log copies/ml] — For PHI-Group HIV RNA at Baseline was measured by Standard Assay. For CHI-Group HIV RNA at Baseline was measured by Single Copy Assay Population: Two Patients of CHI-Group had no single copy measurement.
  log copies/ml
    number analyzed (Participants) | 18 | 22 | 40
    (all) | 0.3 [0.2 to 0.5] | 6.2 [5.3 to 6.9] | NA [NA to NA] — NA=Not available: Baseline HIV RNA was measured with Single copy assay in CHI Group and with Standard Assay in PHI group
Absolute CD4+T cells [Median (Inter-Quartile Range); unit: cells/µl] | 763 [555 to 1065] | 485 [393 to 577] | 570 [453 to 766]
Relative CD4+T cells [Median (Inter-Quartile Range); unit: percent] | 33 [29 to 44] | 24 [17 to 27] | 28 [23 to 36]
CD4+T/CD8+T ratio [Median (Inter-Quartile Range); unit: ratio] — Population: One Patient had no measurement of CD8+T cells .
  ratio
    number analyzed (Participants) | 20 | 21 | 41
    (all) | 0.9 [0.6 to 1.3] | 0.4 [0.3 to 0.6] | 0.6 [0.4 to 0.9]
Absolute CD8+T cells [Median (Inter-Quartile Range); unit: cells/µl] — Population: One Patient had no measurement of CD8+T cells.
  cells/µl
    number analyzed (Participants) | 20 | 21 | 41
    (all) | 864 [782 to 1132] | 1117 [836 to 1615] | 975 [790 to 1268]
Relative CD8+T cells [Median (Inter-Quartile Range); unit: percent] | 39 [34 to 47] | 55 [44 to 64] | 46 [36 to 56]
Absolute CD8+/CD38+ cells [Median (Inter-Quartile Range); unit: cells/µl] — Population: Not all patients had a value for this measurement.
  cells/µl
    number analyzed (Participants) | 15 | 14 | 29
    (all) | 104 [66 to 160] | 872 [506 to 1555] | 204 [104 to 870]
Relative CD8+/CD38+ cells [Median (Inter-Quartile Range); unit: percent] — Population: Not all patients had a value for this measurement.
  percent
    number analyzed (Participants) | 15 | 14 | 29
    (all) | 14 [3.7 to 17] | 89.9 [85. to 94] | 33 [14 to 89]

OUTCOME MEASURES:

1. Primary Outcome: Combined Endpoint Including HIV RNA and HIV DNA
Description: The primary outcome measure (i.e. achievement of 'eradication') is a combined endpoint including cell-associated proviral DNA and plasma HIV RNA and is defined as undetectable cell-associated HIV DNA (copies per 10exp6 PBMC (peripheral blood mononuclear cells) and per 10exp6 CD4 cells) for at least 2 years (measurement by the French ANRS Group) combined with plasma viral load < 50 copies/ml for at least 5 years and undetectable plasma viral load (HIV RNA < 1 copy/ml, 1-copy assay) for at least 2 years.
Time Frame: Screening, month -3 (= pre-baseline only for CHI-patients), baseline, months 1, 3, 6 and then every 6 months until month 84
Population: The efficacy dataset is based on patients who were enrolled in the study, received at least one dose of study drugs and met the inclusion criteria (N=42 patients; efficacy population).
Measure: Count of Participants; unit: Participants
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
Participants | 0 | 0

2. Secondary Outcome: Mean Change in HIV DNA in PBMC (Month 36 and Month 84)
Description: Mean change (CI=95% Confidence Intervall) in HIV DNA copies/10exp6 PBMC (= peripheral blood mononuclear cells) from baseline, to evaluate the decay rates of latently infected cell reservoir.
Time Frame: Change from baseline at months 36 and 84
Population: Data of 42 patients (Efficacy set) at month 36 and 84
Measure: Mean (95% Confidence Interval); unit: log copies/10^6 PBMC
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
log copies/10^6 PBMC
  Month 36: number analyzed (Participants) | 17 | 18
  Month 36 | 0.2 [0.0 to 0.4] | -1.4 [-1.7 to -1.1]
  Month 84: number analyzed (Participants) | 14 | 15
  Month 84 | 0.1 [-0.1 to 0.3] | -1.3 [-1.6 to -1.0]
Statistical Analysis 1: Comparison: CHI-patients; Test type: Other — Changes (within CHI group) in HIV DNA in PBMC from Baseline (BL) will be tested for statistical significance using one-tailed paired t-test or Wilcoxon signed rank test as appropriate on distribution of data at months 36; p = 0.98, t-test, 1 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [0.0 to 0.4]
Statistical Analysis 2: Comparison: PHI-patients; Test type: Other — Changes (within PHI group) in HIV DNA in PBMC from Baseline (BL) will be tested for statistical significance using one-tailed paired t-test or Wilcoxon signed rank test as appropriate on distribution of data at months 36; p < 0.01, t-test, 1 sided; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-1.7 to -1.1]
Statistical Analysis 3: Comparison: CHI-patients; Test type: Other — Changes (within CHI group) in HIV DNA in PBMC from Baseline (BL) will be tested for statistical significance using one-tailed paired t-test or Wilcoxon signed rank test as appropriate on distribution of data at months 84; p = 0.93, t-test, 1 sided; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.1 to 0.3]
Statistical Analysis 4: Comparison: PHI-patients; Test type: Other — Changes (within PHI group) in HIV DNA in PBMC from Baseline (BL) will be tested for statistical significance using one-tailed paired t-test or Wilcoxon signed rank test as appropriate on distribution of data at months 84; p < 0.01, t-test, 1 sided; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-1.6 to -1.0]

3. Secondary Outcome: Mean Change in HIV DNA in CD4+T Cells (Month 36 and Month 84)
Description: Mean change (CI=95% Confidence Intervall) in HIV DNA copies/10exp6 CD4+T cells from baseline, to evaluate the decay rates of latently infected cell reservoir.
Time Frame: Change from baseline at months 36 and 84
Population: Data of 42 patients (Efficacy set) at month 36 and 84
Measure: Mean (95% Confidence Interval); unit: log copies/10^6 PBMC
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
log copies/10^6 PBMC
  Month 36: number analyzed (Participants) | 17 | 18
  Month 36 | 0.2 [0.0 to 0.4] | -1.7 [-2.0 to -1.5]
  Month 84: number analyzed (Participants) | 14 | 15
  Month 84 | 0.2 [-0.0 to 0.3] | -1.7 [-2.0 to -1.4]
Statistical Analysis 1: Comparison: CHI-patients; Test type: Other — Changes (within CHI Group) in HIV DNA in CD4+T cells from Baseline (BL) will be tested for statistical significance using one-tailed paired t-test or Wilcoxon signed rank test as appropriate on distribution of data at month 36; p = 0.99, t-test, 1 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [0.0 to 0.4]
Statistical Analysis 2: Comparison: PHI-patients; Test type: Other — Changes (within PHI Group) in HIV DNA in CD4+T cells from Baseline (BL) will be tested for statistical significance using one-tailed paired t-test or Wilcoxon signed rank test as appropriate on distribution of data at month 36; p < 0.01, t-test, 1 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.0 to -1.5]
Statistical Analysis 3: Comparison: CHI-patients; Test type: Other — Changes (within CHI Group) in HIV DNA in CD4+T cells from Baseline (BL) will be tested for statistical significance using one-tailed paired t-test or Wilcoxon signed rank test as appropriate on distribution of data at month 84; p = 0.97, t-test, 1 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.0 to 0.3]
Statistical Analysis 4: Comparison: PHI-patients; Test type: Other — Changes (within PHI Group) in HIV DNA in CD4+T cells from Baseline (BL) will be tested for statistical significance using one-tailed paired t-test or Wilcoxon signed rank test as appropriate on distribution of data at month 84; p < 0.01, t-test, 1 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.0 to -1.4]

4. Secondary Outcome: HIV RNA <50 Copies/ml (Proportion)
Description: Percentage of patients with Plasma HIV RNA <50 copies/ml at baseline and during follow-up
Time Frame: Baseline and at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Count of Participants; unit: Participants
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
Participants
  Baseline | 20 | 0
  Month1: number analyzed (Participants) | 19 | 22
  Month1 | 18 | 0
  Month 3 | 20 | 12
  Month 6 | 20 | 17
  Month 12 | 20 | 18
  Month 18: number analyzed (Participants) | 20 | 20
  Month 18 | 20 | 19
  Month 24: number analyzed (Participants) | 20 | 20
  Month 24 | 19 | 19
  Month 30: number analyzed (Participants) | 19 | 19
  Month 30 | 19 | 18
  Month 36: number analyzed (Participants) | 19 | 18
  Month 36 | 19 | 18
  Month 42: number analyzed (Participants) | 18 | 18
  Month 42 | 18 | 18
  Month 48: number analyzed (Participants) | 18 | 17
  Month 48 | 17 | 17
  Month 54: number analyzed (Participants) | 18 | 17
  Month 54 | 16 | 17
  Month 60: number analyzed (Participants) | 15 | 17
  Month 60 | 15 | 17
  Month 66: number analyzed (Participants) | 15 | 17
  Month 66 | 15 | 16
  Month 72: number analyzed (Participants) | 15 | 15
  Month 72 | 15 | 14
  Month 78: number analyzed (Participants) | 14 | 15
  Month 78 | 14 | 15
  Month 84: number analyzed (Participants) | 15 | 15
  Month 84 | 14 | 14

5. Secondary Outcome: Median Change in HIV DNA in PBMC Over Time
Description: Median Change from baseline (IQR, interquartile range) in HIV DNA copies/10exp6 PBMC (= peripheral blood mononuclear cells), to evaluate the decay rates of latently infected cell reservoir.
Time Frame: Change from baseline at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: log copies/10^6 PBMC
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
log copies/10^6 PBMC
  Baseline: number analyzed (Participants) | 19 | 22
  Baseline | 0 [0 to 0] | 0 [0 to 0]
  Month 1: number analyzed (Participants) | 18 | 22
  Month 1 | 0.1 [-0.2 to 0.2] | -0.5 [-0.7 to -0.2]
  Month 3: number analyzed (Participants) | 19 | 22
  Month 3 | 0.1 [-0.3 to 0.4] | -0.8 [-1.1 to -0.5]
  Month 6: number analyzed (Participants) | 19 | 21
  Month 6 | 0.1 [-0.2 to 0.3] | -1.0 [-1.3 to -0.7]
  Month 12: number analyzed (Participants) | 19 | 22
  Month 12 | 0.1 [-0.4 to 0.2] | -1.3 [-1.5 to -0.9]
  Month 18: number analyzed (Participants) | 19 | 19
  Month 18 | 0.1 [-0.2 to 0.3] | -1.3 [-1.6 to -1.0]
  Month 24: number analyzed (Participants) | 19 | 20
  Month 24 | 0.2 [-0.1 to 0.4] | -1.4 [-1.7 to -1.2]
  Month 30: number analyzed (Participants) | 18 | 19
  Month 30 | 0.1 [-0.1 to 0.4] | -1.5 [-1.7 to -1.0]
  Month 36: number analyzed (Participants) | 17 | 18
  Month 36 | 0.2 [-0.1 to 0.4] | -1.4 [-1.8 to -1.0]
  Month 42: number analyzed (Participants) | 17 | 17
  Month 42 | 0.1 [0.1 to 0.3] | -1.4 [-1.9 to -1.1]
  Month 48: number analyzed (Participants) | 17 | 22
  Month 48 | 0.2 [-0.0 to 0.4] | -1.6 [-1.7 to -1.4]
  Month 54: number analyzed (Participants) | 16 | 16
  Month 54 | 0.2 [0 to 0.4] | -1.5 [-1.8 to -1.1]
  Month 60: number analyzed (Participants) | 14 | 17
  Month 60 | 0.1 [-0.0 to 0.4] | -1.6 [-1.7 to -1.2]
  Month 66: number analyzed (Participants) | 14 | 16
  Month 66 | 0.1 [-0.0 to 0.4] | -1.5 [-2.0 to -1.0]
  Month 72: number analyzed (Participants) | 14 | 16
  Month 72 | 0.2 [-0.1 to 0.4] | -1.5 [-1.7 to -1.3]
  Month 78: number analyzed (Participants) | 12 | 15
  Month 78 | 0.2 [0.0 to 0.6] | -1.6 [-2.2 to -0.9]
  Month 84: number analyzed (Participants) | 14 | 15
  Month 84 | 0.0 [-0.1 to 0.4] | -1.4 [-1.8 to -0.8]

6. Secondary Outcome: Median Change in HIV DNA in CD4+T Cells Over Time
Description: Median Change from baseline (IQR, interquartile range) in HIV DNA in CD4+T cells, to evaluate the decay rates of latently infected cell reservoir.
Time Frame: Change from baseline at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: log copies/10^6 CD4+T cells
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
log copies/10^6 CD4+T cells
  Baseline: number analyzed (Participants) | 19 | 22
  Baseline | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 1: number analyzed (Participants) | 18 | 22
  Month 1 | 0.1 [-0.2 to 0.3] | -0.7 [-0.9 to -0.4]
  Month 3: number analyzed (Participants) | 19 | 22
  Month 3 | 0.1 [-0.3 to 0.4] | -1.1 [-1.3 to -0.8]
  Month 6: number analyzed (Participants) | 19 | 21
  Month 6 | 0.1 [-0.2 to 0.4] | -1.3 [-1.6 to -0.9]
  Month 12: number analyzed (Participants) | 19 | 22
  Month 12 | 0.1 [-0.3 to 0.2] | -1.6 [-1.8 to -1.2]
  Month 18: number analyzed (Participants) | 19 | 19
  Month 18 | 0.1 [-0.1 to 0.3] | -1.6 [-1.8 to -1.3]
  Month 24: number analyzed (Participants) | 19 | 20
  Month 24 | 0.3 [0.1 to 0.4] | -1.7 [-2.0 to -1.5]
  Month 30: number analyzed (Participants) | 18 | 19
  Month 30 | 0.2 [-0.1 to 0.3] | -1.7 [-2.0 to -1.3]
  Month 36: number analyzed (Participants) | 17 | 18
  Month 36 | 0.1 [-0.0 to 0.4] | -1.7 [-2.1 to -1.3]
  Month 42: number analyzed (Participants) | 17 | 17
  Month 42 | 0.1 [0.1 to 0.3] | -1.7 [-2.0 to -1.5]
  Month 48: number analyzed (Participants) | 17 | 17
  Month 48 | 0.2 [0.1 to 0.3] | -1.9 [-2.1 to -1.5]
  Month 54: number analyzed (Participants) | 16 | 16
  Month 54 | 0.2 [0.0 to 0.4] | -1.7 [-2.1 to -1.5]
  Month 60: number analyzed (Participants) | 14 | 17
  Month 60 | 0.1 [-0.0 to 0.4] | -1.8 [-1.9 to -1.6]
  Month 66: number analyzed (Participants) | 14 | 16
  Month 66 | 0.1 [-0.0 to 0.4] | -1.7 [-2.3 to -1.5]
  Month 72: number analyzed (Participants) | 14 | 16
  Month 72 | 0.2 [-0.0 to 0.3] | -1.8 [-2.1 to -1.6]
  Month 78: number analyzed (Participants) | 12 | 15
  Month 78 | 0.2 [0.1 to 0.5] | -2.0 [-2.4 to -1.5]
  Month 84: number analyzed (Participants) | 14 | 15
  Month 84 | 0.1 [-0.1 to 0.4] | -1.7 [-2.2 to -1.4]

7. Secondary Outcome: Median Change in CD4+T Cells Over Time
Description: Median Change from baseline (IQR, interquartile range) in CD4+T cells/µl.
Time Frame: Change from baseline at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: cells/µl
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
cells/µl
  Baseline | 0 [0 to 0] | 0 [0 to 0]
  Month 1: number analyzed (Participants) | 19 | 22
  Month 1 | 10 [-54.0 to 159.0] | 272.0 [158.0 to 413.0]
  Month 3 | 22 [-45.0 to 109.0] | 425.0 [173.0 to 506.0]
  Month 6 | 51.5 [-71.5 to 111.0] | 344.0 [169.0 to 566.0]
  Month 12 | 17 [-89.0 to 103.5] | 496.0 [222.0 to 619.0]
  Month 18: number analyzed (Participants) | 20 | 20
  Month 18 | 75.5 [-3.0 to 190.5] | 447.0 [220.0 to 692.0]
  Month 24: number analyzed (Participants) | 20 | 20
  Month 24 | 52 [-39.5 to 116.5] | 423.0 [239.5 to 792.5]
  Month 30: number analyzed (Participants) | 19 | 19
  Month 30 | 80 [-37.0 to 132.0] | 420.0 [224.0 to 751.0]
  Month 36: number analyzed (Participants) | 19 | 18
  Month 36 | 45 [-19.0 to 150.0] | 395.5 [192.0 to 678.0]
  Month 42: number analyzed (Participants) | 18 | 18
  Month 42 | 36.5 [-41.0 to 148.0] | 365.0 [228.0 to 523.0]
  Month 48: number analyzed (Participants) | 18 | 17
  Month 48 | 48.5 [10.0 to 128.0] | 404.0 [254.0 to 723.0]
  Month 54: number analyzed (Participants) | 18 | 17
  Month 54 | 80 [-122.0 to 162.0] | 484.0 [302.0 to 646.0]
  Month 60: number analyzed (Participants) | 15 | 17
  Month 60 | 60 [-78.0 to 207.0] | 383.0 [263.0 to 724.0]
  Month 66: number analyzed (Participants) | 15 | 17
  Month 66 | 70 [-87.0 to 141.0] | 413.0 [287.0 to 565.0]
  Month 72: number analyzed (Participants) | 15 | 16
  Month 72 | 99 [-40.0 to 215.0] | 476.5 [356.0 to 641.5]
  Month 78: number analyzed (Participants) | 14 | 15
  Month 78 | 32 [-55.0 to 275.0] | 389.0 [184.0 to 647.0]
  Month 84: number analyzed (Participants) | 15 | 15
  Month 84 | 49 [-142.0 to 180.0] | 457.0 [242.0 to 578.0]

8. Secondary Outcome: Median Change in Relative CD4+T Cells Over Time
Description: Median Change from baseline (IQR, interquartile range) in relative CD4+T cells/µl.
Time Frame: Change from baseline at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: percentage of Lymphocytes
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
percentage of Lymphocytes
  Baseline | 0 [0 to 0] | 0 [0 to 0]
  Month 1: number analyzed (Participants) | 19 | 22
  Month 1 | -1.0 [-3.0 to 0.0] | 13.5 [9.0 to 17.0]
  Month 3 | -1.8 [-3.0 to 0.8] | 14.0 [9.0 to 19.0]
  Month 6 | -1.5 [-3.5 to 0.8] | 18.5 [10.0 to 23.0]
  Month 12 | -1.3 [-4.5 to 1.0] | 17.5 [11.0 to 25.0]
  Month 18: number analyzed (Participants) | 20 | 20
  Month 18 | -2.0 [-6.0 to 0.0] | 18.0 [13.0 to 23.5]
  Month 24: number analyzed (Participants) | 20 | 20
  Month 24 | -2.5 [-4.5 to 1.8] | 18.5 [14.0 to 24.0]
  Month 30: number analyzed (Participants) | 19 | 19
  Month 30 | -1.6 [-4.0 to 0.0] | 16.0 [13.0 to 27.0]
  Month 36: number analyzed (Participants) | 19 | 18
  Month 36 | -0.6 [-4.0 to 2.0] | 19.0 [13.0 to 25.0]
  Month 42: number analyzed (Participants) | 18 | 18
  Month 42 | -0.5 [-5.0 to 3.0] | 18.5 [12.0 to 25.6]
  Month 48: number analyzed (Participants) | 18 | 17
  Month 48 | -0.5 [-5.0 to 2.0] | 17.0 [10.0 to 27.0]
  Month 54: number analyzed (Participants) | 18 | 17
  Month 54 | 0.5 [-6.7 to 2.0] | 20.0 [13.0 to 27.1]
  Month 60: number analyzed (Participants) | 15 | 17
  Month 60 | 2.0 [-3.0 to 4.0] | 18.0 [12.0 to 26.0]
  Month 66: number analyzed (Participants) | 15 | 17
  Month 66 | 1.0 [-5.0 to 4.0] | 17.0 [12.0 to 26.9]
  Month 72: number analyzed (Participants) | 15 | 16
  Month 72 | 0.0 [-3.0 to 7.0] | 18.2 [11.0 to 25.5]
  Month 78: number analyzed (Participants) | 14 | 15
  Month 78 | 0.0 [-5.0 to 3.0] | 20.0 [15.0 to 24.7]
  Month 84: number analyzed (Participants) | 15 | 15
  Month 84 | 0.0 [-6.1 to 5.0] | 22.0 [11.0 to 31.0]

9. Secondary Outcome: Median Change in CD4+/CD8+ Ratio Over Time
Description: Median change in CD4+/ CD8+ ratio at baseline (IQR, interquartile range) and during follow-up
Time Frame: Change form Baseline at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
ratio
  Baseline: number analyzed (Participants) | 20 | 21
  Baseline | 0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 1: number analyzed (Participants) | 19 | 21
  Month 1 | -0.0 [-0.2 to 0.0] | 0.5 [0.3 to 0.8]
  Month 3: number analyzed (Participants) | 20 | 21
  Month 3 | -0.1 [-0.2 to 0.0] | 0.5 [0.4 to 1.0]
  Month 6: number analyzed (Participants) | 20 | 21
  Month 6 | -0.1 [-0.1 to 0.0] | 0.7 [0.6 to 1.0]
  Month 12: number analyzed (Participants) | 20 | 21
  Month 12 | -0.1 [-0.2 to 0.1] | 0.8 [0.7 to 1.1]
  Month 18: number analyzed (Participants) | 20 | 19
  Month 18 | -0.1 [-0.3 to 0.0] | 0.8 [0.8 to 1.1]
  Month 24: number analyzed (Participants) | 20 | 19
  Month 24 | -0.1 [-0.2 to 0.0] | 0.9 [0.8 to 1.3]
  Month 30: number analyzed (Participants) | 19 | 18
  Month 30 | -0.1 [-0.3 to 0.0] | 0.8 [0.7 to 1.2]
  Month 36: number analyzed (Participants) | 19 | 17
  Month 36 | -0.0 [-0.3 to 0.1] | 1.0 [0.8 to 1.2]
  Month 42: number analyzed (Participants) | 18 | 16
  Month 42 | -0.1 [-0.2 to 0.0] | 1.0 [0.7 to 1.2]
  Month 48: number analyzed (Participants) | 18 | 16
  Month 48 | -0.0 [-0.1 to 0.1] | 0.9 [0.7 to 1.2]
  Month 54: number analyzed (Participants) | 18 | 16
  Month 54 | 0.0 [-0.1 to 0.1] | 1.1 [0.8 to 1.2]
  Month 60: number analyzed (Participants) | 15 | 16
  Month 60 | 0.1 [-0.1 to 0.3] | 0.9 [0.8 to 1.4]
  Month 66: number analyzed (Participants) | 15 | 16
  Month 66 | 0.1 [-0.1 to 0.1] | 0.9 [0.7 to 1.2]
  Month 72: number analyzed (Participants) | 14 | 16
  Month 72 | 0 [-0.2 to 0.3] | 0.8 [0.6 to 1.4]
  Month 78: number analyzed (Participants) | 14 | 14
  Month 78 | 0 [-0.1 to 0.1] | 0.9 [0.8 to 1.0]
  Month 84: number analyzed (Participants) | 15 | 14
  Month 84 | 0.1 [-0.2 to 0.1] | 0.9 [0.7 to 1.8]

10. Secondary Outcome: Median Change in CD8+T Cells Over Time
Description: Median Change from baseline (IQR, interquartile range) in CD8+T cells/µl.
Time Frame: Change from baseline at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: cells/µl
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
cells/µl
  Baseline: number analyzed (Participants) | 20 | 21
  Baseline | 0 [0 to 0] | 0 [0 to 0]
  Month 1: number analyzed (Participants) | 19 | 21
  Month 1 | 64.0 [-63.0 to 213.0] | -405.0 [-822.0 to -43.0]
  Month 3: number analyzed (Participants) | 20 | 21
  Month 3 | 114.5 [-24.0 to 236.5] | -375.0 [-1021.0 to -42.0]
  Month 6: number analyzed (Participants) | 20 | 21
  Month 6 | 141.0 [-32.0 to 215.0] | -505.0 [-726.0 to -153.0]
  Month 12: number analyzed (Participants) | 20 | 21
  Month 12 | 32.0 [-118.5 to 238.0] | -394.0 [-880.0 to -249.0]
  Month 18: number analyzed (Participants) | 20 | 19
  Month 18 | 224.0 [41.5 to 455.0] | -377.0 [-863.0 to -216.0]
  Month 24: number analyzed (Participants) | 20 | 19
  Month 24 | 167.0 [3.0 to 357.0] | -376.0 [-881.0 to -249.0]
  Month 30: number analyzed (Participants) | 19 | 18
  Month 30 | 220.0 [-49.0 to 420.0] | -406.0 [-1007.0 to -196.0]
  Month 36: number analyzed (Participants) | 19 | 17
  Month 36 | 170.0 [41.0 to 350.0] | -456.0 [-826.0 to -310.0]
  Month 42: number analyzed (Participants) | 18 | 16
  Month 42 | 170.0 [-22.0 to 298.0] | -460.5 [-1022.5 to -207.0]
  Month 48: number analyzed (Participants) | 18 | 16
  Month 48 | 80.5 [21.0 to 261.0] | -562.0 [-1182.5 to -98.5]
  Month 54: number analyzed (Participants) | 18 | 16
  Month 54 | 88.5 [-140.0 to 246.0] | -507.0 [-1220.0 to -233.5]
  Month 60: number analyzed (Participants) | 15 | 16
  Month 60 | 123.0 [-237.0 to 325.0] | -418.0 [-1305.0 to -252.0]
  Month 66: number analyzed (Participants) | 15 | 16
  Month 66 | 33.0 [-40.0 to 520.0] | -467.5 [-1271.5 to -267.5]
  Month 72: number analyzed (Participants) | 14 | 16
  Month 72 | 123.0 [-54.0 to 291.0] | -446.0 [-1237.0 to -97.5]
  Month 78: number analyzed (Participants) | 14 | 14
  Month 78 | 212.5 [0.0 to 500.0] | -494.0 [-1769.0 to -147.0]
  Month 84: number analyzed (Participants) | 15 | 14
  Month 84 | 35.0 [-161.0 to 143.0] | -443.0 [-1670.0 to -185.0]

11. Secondary Outcome: Median Change in CD8+CD38+T Cells Over Time
Description: Median Change from baseline (IQR, interquartile range) in CD8+CD38+T cells/µl.
Time Frame: Change from baseline at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: cells/µl
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
cells/µl
  Baseline: number analyzed (Participants) | 15 | 14
  Baseline | 0 [0 to 0] | 0 [0 to 0]
  Month 1: number analyzed (Participants) | 13 | 13
  Month 1 | 19.0 [0.0 to 61.0] | -488.0 [-757.0 to -192.0]
  Month 3: number analyzed (Participants) | 13 | 12
  Month 3 | 51.9 [-1.0 to 114.0] | -776.5 [-1726.5 to -451.0]
  Month 6: number analyzed (Participants) | 13 | 14
  Month 6 | 24.0 [3.0 to 97.0] | -646.5 [-1474.0 to -484.0]
  Month 12: number analyzed (Participants) | 13 | 10
  Month 12 | 32.0 [-3.0 to 51.0] | -897.0 [-1478.0 to -583.0]
  Month 18: number analyzed (Participants) | 14 | 10
  Month 18 | 50.5 [-17.0 to 125.0] | -744.0 [-1394.0 to -464.0]
  Month 24: number analyzed (Participants) | 15 | 11
  Month 24 | 2.0 [-33.0 to 49.0] | -786.0 [-2086.0 to -456.0]
  Month 30: number analyzed (Participants) | 11 | 11
  Month 30 | 4.0 [-36.0 to 64.0] | -772.0 [-2154.0 to -467.0]
  Month 36: number analyzed (Participants) | 13 | 9
  Month 36 | 11.0 [-32.0 to 73.0] | -1077.0 [-2170.0 to -500.0]
  Month 42: number analyzed (Participants) | 13 | 10
  Month 42 | -15.0 [-48.0 to 5.0] | -726.0 [-1429.0 to -467.0]
  Month 48: number analyzed (Participants) | 11 | 9
  Month 48 | -2.0 [-53.0 to 243.0] | -1070.0 [-2149.0 to -468.2]
  Month 54: number analyzed (Participants) | 13 | 11
  Month 54 | -10.0 [-62.0 to 72.0] | -729.0 [-1446.0 to -466.0]
  Month 60: number analyzed (Participants) | 11 | 10
  Month 60 | -13.0 [-42.0 to 115.0] | -752.0 [-1401.0 to -452.0]
  Month 66: number analyzed (Participants) | 11 | 11
  Month 66 | -22.1 [-71.0 to 72.0] | -777.0 [-1431.0 to -469.0]
  Month 72: number analyzed (Participants) | 10 | 11
  Month 72 | 3.5 [-57.0 to 44.0] | -810.0 [-1438.0 to -485.9]
  Month 78: number analyzed (Participants) | 9 | 9
  Month 78 | 31.0 [-73.0 to 77.0] | -730.0 [-1523.0 to -474.2]
  Month 84: number analyzed (Participants) | 10 | 8
  Month 84 | -22.5 [-82.0 to 17.9] | -1201.5 [-2454.0 to -621.0]

12. Secondary Outcome: Absolute HIV DNA in PBMC
Description: Absolute HIV DNA in PBMC (= peripheral blood mononuclear cells) from baseline (Median; IQR, interquartile range), to quantify the cell-associated latently infected reservoir size by visit and treatment Group.
Time Frame: Baseline and at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: log copies/10^6 PBMC
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
log copies/10^6 PBMC
  Baseline: number analyzed (Participants) | 19 | 22
  Baseline | 2.5 [2.0 to 2.7] | 3.6 [3.5 to 3.8]
  Month 1: number analyzed (Participants) | 18 | 22
  Month 1 | 2.4 [2.2 to 2.7] | 3.1 [2.9 to 3.5]
  Month 3 | 2.6 [2.2 to 2.7] | 2.7 [2.6 to 3.1]
  Month 6: number analyzed (Participants) | 20 | 21
  Month 6 | 2.6 [2.3 to 2.7] | 2.5 [2.3 to 2.8]
  Month 12 | 2.4 [2.2 to 2.6] | 2.2 [2.0 to 2.7]
  Month 18: number analyzed (Participants) | 20 | 19
  Month 18 | 2.6 [2.3 to 2.8] | 2.2 [2.0 to 2.6]
  Month 24: number analyzed (Participants) | 20 | 20
  Month 24 | 2.6 [2.4 to 2.9] | 2.1 [1.9 to 2.3]
  Month 30: number analyzed (Participants) | 19 | 19
  Month 30 | 2.7 [2.2 to 2.8] | 2.2 [1.9 to 2.5]
  Month 36: number analyzed (Participants) | 17 | 18
  Month 36 | 2.7 [2.5 to 2.8] | 2.2 [1.9 to 2.3]
  Month 42: number analyzed (Participants) | 17 | 17
  Month 42 | 2.6 [2.4 to 2.8] | 2.0 [1.7 to 2.4]
  Month 48: number analyzed (Participants) | 18 | 17
  Month 48 | 2.6 [2.4 to 2.8] | 2.1 [1.8 to 2.1]
  Month 54: number analyzed (Participants) | 17 | 17
  Month 54 | 2.6 [2.4 to 2.6] | 2.1 [2.0 to 2.2]
  Month 60: number analyzed (Participants) | 15 | 17
  Month 60 | 2.5 [2.3 to 2.8] | 2.1 [1.9 to 2.2]
  Month 66: number analyzed (Participants) | 15 | 16
  Month 66 | 2.6 [2.4 to 2.8] | 1.9 [1.7 to 2.2]
  Month 72: number analyzed (Participants) | 15 | 16
  Month 72 | 2.6 [2.4 to 2.8] | 1.9 [1.8 to 2.2]
  Month 78: number analyzed (Participants) | 13 | 15
  Month 78 | 2.6 [2.4 to 2.8] | 2.0 [1.7 to 2.6]
  Month 84: number analyzed (Participants) | 15 | 15
  Month 84 | 2.4 [2.4 to 2.8] | 2.3 [2.0 to 2.6]

13. Secondary Outcome: Absolute HIV DNA in CD4+T Cells
Description: Absolute HIV DNA in CD4+T cells from baseline (Median; IQR, interquartile range), to quantify the cell-associated latently infected reservoir size by visit and treatment Group.
Time Frame: Baseline and at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: log copies/10^6 CD4+T cells
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
log copies/10^6 CD4+T cells
  Baseline: number analyzed (Participants) | 19 | 22
  Baseline | 3.0 [2.6 to 3.3] | 4.4 [4.1 to 4.6]
  Month1: number analyzed (Participants) | 18 | 22
  Month1 | 3.0 [2.8 to 3.4] | 3.6 [3.3 to 4.0]
  Month 3 | 3.1 [2.9 to 3.3] | 3.2 [3.0 to 3.6]
  Month 6: number analyzed (Participants) | 20 | 21
  Month 6 | 3.1 [2.7 to 3.2] | 3.0 [2.8 to 3.2]
  Month 12 | 3.0 [2.8 to 3.2] | 2.6 [2.5 to 3.1]
  Month 18: number analyzed (Participants) | 20 | 19
  Month 18 | 3.2 [2.9 to 3.3] | 2.7 [2.3 to 3.0]
  Month 24: number analyzed (Participants) | 20 | 20
  Month 24 | 3.3 [3.0 to 3.5] | 2.6 [2.3 to 2.8]
  Month 30: number analyzed (Participants) | 19 | 19
  Month 30 | 3.2 [2.8 to 3.3] | 2.6 [2.4 to 2.9]
  Month 36: number analyzed (Participants) | 17 | 18
  Month 36 | 3.2 [3.0 to 3.4] | 2.7 [2.4 to 2.8]
  Month 42: number analyzed (Participants) | 17 | 17
  Month 42 | 3.2 [2.9 to 3.4] | 2.5 [2.1 to 2.8]
  Month 48: number analyzed (Participants) | 18 | 17
  Month 48 | 3.2 [3.0 to 3.3] | 2.5 [2.4 to 2.7]
  Month 54: number analyzed (Participants) | 17 | 16
  Month 54 | 3.1 [2.9 to 3.2] | 2.5 [2.4 to 2.7]
  Month 60: number analyzed (Participants) | 15 | 17
  Month 60 | 3.1 [2.8 to 3.4] | 2.5 [2.3 to 2.7]
  Month 66: number analyzed (Participants) | 15 | 16
  Month 66 | 3.3 [3.0 to 3.4] | 2.3 [2.2 to 2.7]
  Month 72: number analyzed (Participants) | 15 | 16
  Month 72 | 3.1 [2.9 to 3.4] | 2.4 [2.2 to 2.7]
  Month 78: number analyzed (Participants) | 13 | 15
  Month 78 | 3.3 [3.1 to 3.4] | 2.6 [2.2 to 3.1]
  Month 84: number analyzed (Participants) | 15 | 15
  Month 84 | 3.1 [2.9 to 3.4] | 2.7 [2.3 to 3.1]

14. Secondary Outcome: Absolute CD4+T Cells
Description: Median CD4+T cells/µl at baseline (IQR, interquartile range) and during follow-up
Time Frame: Baseline and at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: cells/µl
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
cells/µl
  Baseline | 762.5 [554.5 to 1065.0] | 484.5 [393.0 to 577.0]
  Month 1 | 653.0 [534.0 to 1098.0] | 796.5 [654.0 to 915.0]
  Month 3 | 801.5 [596.5 to 919.5] | 801.0 [599.0 to 1116.0]
  Month 6 | 798.0 [588.5 to 975.5] | 854.5 [685.0 to 983.0]
  Month 12 | 749.0 [567.0 to 920.5] | 943.5 [688.0 to 1071.0]
  Month 18 | 815.5 [615.0 to 1200.5] | 981.5 [666.0 to 1175.5]
  Month 24 | 766.5 [593.5 to 1041.5] | 927.5 [721.0 to 1303.0]
  Month 30 | 703.0 [537.0 to 1110.0] | 840.0 [641.0 to 1208.0]
  Month 36 | 827.0 [565.0 to 1145.0] | 915.5 [638.0 to 1179.0]
  Month 42 | 721.5 [590.0 to 997.0] | 827.5 [708.0 to 1157.0]
  Month 48 | 822.0 [589.0 to 1123.0] | 945.0 [606.0 to 1169.0]
  Month 54 | 879.5 [570.0 to 927.0] | 880.0 [658.0 to 1210.0]
  Month 60 | 880.0 [744.0 to 1021.0] | 877.0 [722.0 to 1139.0]
  Month 66 | 749.0 [620.0 to 1014.0] | 977.0 [685.0 to 1133.0]
  Month 72 | 843.0 [629.0 to 1052.0] | 940.0 [806.5 to 1169.0]
  Month 78 | 798.0 [618.0 to 940.0] | 802.0 [577.0 to 1112.0]
  Month 84 | 733.0 [545.0 to 964.0] | 938.0 [739.0 to 1164.0]

15. Secondary Outcome: Relative CD4+T Cells
Description: Median relative CD4+T cells/µl at baseline (IQR, interquartile range) and during follow-up
Time Frame: Baseline and at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: percentage of Lymphocytes
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
percentage of Lymphocytes
  Baseline | 32.5 [28.5 to 43.5] | 24.0 [17.0 to 27.0]
  Month 1: number analyzed (Participants) | 19 | 22
  Month 1 | 32.0 [28.0 to 41.0] | 34.0 [32.0 to 40.0]
  Month 3 | 31.0 [28.0 to 41.0] | 35.5 [31.0 to 42.0]
  Month 6 | 35.0 [25.5 to 40.1] | 38.5 [36.0 to 45.0]
  Month 12 | 30.5 [26.0 to 40.0] | 40.0 [38.0 to 43.0]
  Month 18 | 31.0 [26.5 to 38.0] | 40.0 [37.5 to 44.0]
  Month 24: number analyzed (Participants) | 20 | 20
  Month 24 | 30.0 [26.5 to 39.5] | 40.0 [37.0 to 45.5]
  Month 30: number analyzed (Participants) | 19 | 19
  Month 30 | 31.5 [29.0 to 42.0] | 40.0 [37.0 to 43.0]
  Month 36: number analyzed (Participants) | 19 | 18
  Month 36 | 33.0 [28.0 to 43.6] | 41.0 [38.0 to 46.0]
  Month 42: number analyzed (Participants) | 18 | 18
  Month 42 | 32.0 [26.0 to 40.0] | 41.0 [38.0 to 47.0]
  Month 48: number analyzed (Participants) | 18 | 17
  Month 48 | 33.5 [26.0 to 39.0] | 39.0 [36.9 to 45.0]
  Month 54: number analyzed (Participants) | 18 | 17
  Month 54 | 33.0 [28.0 to 43.0] | 42.0 [38.0 to 46.0]
  Month 60: number analyzed (Participants) | 15 | 17
  Month 60 | 34.0 [27.0 to 42.0] | 40.7 [40.0 to 44.0]
  Month 66: number analyzed (Participants) | 15 | 17
  Month 66 | 31.0 [24.0 to 35.0] | 40.0 [38.0 to 46.0]
  Month 72: number analyzed (Participants) | 15 | 16
  Month 72 | 35.0 [23.0 to 40.0] | 41.5 [37.0 to 45.5]
  Month 78: number analyzed (Participants) | 14 | 15
  Month 78 | 31.5 [22.0 to 34.0] | 40.0 [37.0 to 47.0]
  Month 84: number analyzed (Participants) | 15 | 15
  Month 84 | 32.0 [24.0 to 39.0] | 43.0 [36.6 to 48.0]

16. Secondary Outcome: CD4+/CD8+ Ratio
Description: Median CD4+/CD8+ ratio at baseline (IQR, interquartile range) and during follow-up
Time Frame: Baseline and at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
ratio
  Baseline | 0.9 [0.6 to 1.3] | 0.4 [0.3 to 0.6]
  Month 1: number analyzed (Participants) | 19 | 22
  Month 1 | 0.9 [0.6 to 1.2] | 1.0 [0.7 to 1.2]
  Month 3 | 0.8 [0.6 to 1.1] | 1.0 [0.8 to 1.7]
  Month 6 | 0.8 [0.6 to 1.1] | 1.2 [1.0 to 1.6]
  Month 12 | 0.7 [0.6 to 1.1] | 1.3 [1.2 to 1.8]
  Month 18: number analyzed (Participants) | 20 | 20
  Month 18 | 0.7 [0.6 to 1.0] | 1.3 [1.1 to 1.8]
  Month 24: number analyzed (Participants) | 20 | 20
  Month 24 | 0.8 [0.6 to 1.0] | 1.5 [1.1 to 1.8]
  Month 30: number analyzed (Participants) | 19 | 19
  Month 30 | 0.7 [0.5 to 1.2] | 1.3 [1.1 to 1.8]
  Month 36: number analyzed (Participants) | 19 | 18
  Month 36 | 0.8 [0.6 to 1.1] | 1.3 [1.1 to 1.9]
  Month 42: number analyzed (Participants) | 18 | 17
  Month 42 | 0.8 [0.5 to 1.1] | 1.3 [1.1 to 1.9]
  Month 48: number analyzed (Participants) | 18 | 17
  Month 48 | 0.8 [0.6 to 1.1] | 1.5 [1.1 to 1.8]
  Month 54: number analyzed (Participants) | 18 | 17
  Month 54 | 0.9 [0.7 to 1.4] | 1.5 [1.1 to 2.0]
  Month 60: number analyzed (Participants) | 15 | 17
  Month 60 | 0.9 [0.6 to 1.3] | 1.4 [1.1 to 1.8]
  Month 66: number analyzed (Participants) | 15 | 17
  Month 66 | 0.9 [0.5 to 1.0] | 1.3 [1.2 to 1.8]
  Month 72: number analyzed (Participants) | 14 | 16
  Month 72 | 0.8 [0.5 to 1.2] | 1.5 [1.1 to 1.8]
  Month 78: number analyzed (Participants) | 14 | 15
  Month 78 | 0.7 [0.5 to 1.0] | 1.4 [1.0 to 1.8]
  Month 84: number analyzed (Participants) | 15 | 15
  Month 84 | 0.7 [0.5 to 1.0] | 1.4 [1.0 to 2.1]

17. Secondary Outcome: Absolute CD8+T Cells
Description: Median CD8+T cells/µl at baseline (IQR, interquartile range) and during follow-up
Time Frame: Baseline and at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: cells/µl
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
cells/µl
  Baseline: number analyzed (Participants) | 20 | 21
  Baseline | 864.0 [782.0 to 1132.0] | 1117.0 [836.0 to 1615.0]
  Month 1: number analyzed (Participants) | 19 | 22
  Month 1 | 949.0 [640.0 to 1220.0] | 806.0 [544.0 to 1014.0]
  Month 3 | 904.0 [841.5 to 1320.0] | 768.5 [567.0 to 1147.0]
  Month 6 | 980.0 [744.0 to 1233.0] | 705.0 [512.0 to 951.0]
  Month 12 | 1031.0 [649.5 to 1249.5] | 721.5 [483.0 to 897.0]
  Month 18: number analyzed (Participants) | 20 | 20
  Month 18 | 1193.5 [893.0 to 1465.5] | 692.0 [508.5 to 934.0]
  Month 24: number analyzed (Participants) | 20 | 20
  Month 24 | 1133.5 [889.0 to 1320.0] | 684.0 [528.0 to 937.5]
  Month 30: number analyzed (Participants) | 19 | 19
  Month 30 | 1103.0 [725.0 to 1468.0] | 677.0 [488.0 to 936.0]
  Month 36: number analyzed (Participants) | 19 | 18
  Month 36 | 1010.0 [858.0 to 1330.0] | 589.0 [466.0 to 851.0]
  Month 42: number analyzed (Participants) | 18 | 17
  Month 42 | 1066.0 [881.0 to 1363.0] | 630.0 [543.0 to 710.0]
  Month 48: number analyzed (Participants) | 18 | 17
  Month 48 | 975.0 [709.0 to 1255.0] | 669.0 [473.0 to 767.0]
  Month 54: number analyzed (Participants) | 18 | 17
  Month 54 | 975.0 [672.0 to 1300.0] | 625.0 [506.0 to 746.0]
  Month 60: number analyzed (Participants) | 15 | 17
  Month 60 | 1002.0 [657.0 to 1242.0] | 650.0 [542.0 to 828.0]
  Month 66: number analyzed (Participants) | 15 | 17
  Month 66 | 1072.0 [807.0 to 1368.0] | 630.0 [464.0 to 835.0]
  Month 72: number analyzed (Participants) | 14 | 16
  Month 72 | 1062.5 [720.0 to 1473.0] | 695.0 [516.0 to 833.5]
  Month 78: number analyzed (Participants) | 14 | 15
  Month 78 | 1196.5 [1008.0 to 1615.0] | 592.0 [412.0 to 869.0]
  Month 84: number analyzed (Participants) | 15 | 15
  Month 84 | 1000.0 [820.0 to 1189.0] | 692.0 [511.0 to 825.0]

18. Secondary Outcome: Absolute CD8+CD38+T Cells
Description: Median CD8+CD38+T cells/µl at baseline (IQR, interquartile range) and during follow-up
Time Frame: Baseline and at months 1, 3, 6 and then every 6 months until month 84
Population: Data of 42 patients (Efficacy set)
Measure: Median (Inter-Quartile Range); unit: cells/µl
Arm/Group | CHI-patients | PHI-patients
Number analyzed (Participants) | 20 | 22
cells/µl
  Baseline: number analyzed (Participants) | 15 | 14
  Baseline | 104.0 [66.0 to 160.0] | 871.5 [506.0 to 1555.0]
  Month 1: number analyzed (Participants) | 16 | 15
  Month 1 | 113.5 [85.5 to 191.5] | 406.0 [192.0 to 696.0]
  Month 3: number analyzed (Participants) | 16 | 17
  Month 3 | 165.5 [99.5 to 282.5] | 202.0 [149.0 to 322.0]
  Month 6: number analyzed (Participants) | 16 | 21
  Month 6 | 182.5 [113.5 to 234.0] | 151.0 [74.0 to 184.0]
  Month 12: number analyzed (Participants) | 16 | 17
  Month 12 | 161.0 [111.0 to 204.5] | 106.0 [56.0 to 143.0]
  19Month 18: number analyzed (Participants) | 18 | 15
  19Month 18 | 203.5 [77.0 to 280.0] | 97.0 [67.0 to 175.0]
  Month 24: number analyzed (Participants) | 19 | 19
  Month 24 | 129.0 [74.0 to 241.0] | 71.0 [28.0 to 171.0]
  Month 30: number analyzed (Participants) | 15 | 17
  Month 30 | 128.0 [72.0 to 199.0] | 86.0 [69.0 to 135.0]
  Month 36: number analyzed (Participants) | 17 | 15
  Month 36 | 163.0 [63.0 to 191.0] | 79.0 [12.0 to 121.0]
  Month 42: number analyzed (Participants) | 18 | 17
  Month 42 | 144.5 [47.0 to 210.0] | 102.0 [42.0 to 121.0]
  Month 48: number analyzed (Participants) | 16 | 14
  Month 48 | 147.0 [62.0 to 274.5] | 78.0 [40.0 to 132.0]
  Month 54: number analyzed (Participants) | 18 | 17
  Month 54 | 80.0 [50.0 to 208.0] | 81.0 [25.0 to 140.0]
  Month 60: number analyzed (Participants) | 15 | 14
  Month 60 | 110.0 [40.0 to 180.0] | 69.0 [39.0 to 109.0]
  Month 66: number analyzed (Participants) | 15 | 15
  Month 66 | 100.0 [33.0 to 195.0] | 69.0 [31.0 to 136.0]
  Month 72: number analyzed (Participants) | 15 | 14
  Month 72 | 110.0 [46.0 to 217.0] | 53.0 [33.0 to 120.4]
  Month 78: number analyzed (Participants) | 13 | 13
  Month 78 | 134.0 [80.0 to 330.0] | 60.0 [23.0 to 125.0]
  Month 84: number analyzed (Participants) | 14 | 13
  Month 84 | 120.0 [48.0 to 170.0] | 64.0 [37.0 to 156.0]

ADVERSE EVENTS:
Time Frame: Adverse events per Patient were collected at the conducted half-yearly study visits, beginnig on individual study start up to the end of study (Month 84) or up to premature discontinuation. In case of premature discontinuation the adverse events occurring during post-follow-up observation period are also included in this report.
Description: The safety dataset (safety population) is based on all patients enrolled in the study and having received at least one dose of study drugs, i.e. 42 eligible patients enrolled in the study (=efficacy dataset), and in addition 5 patients with primary HIV infection, who immediately started on study drugs (as defined by the study protocol) but turned out to be screening failures upon laboratory findings. The count of patients differed between both datasets (safety dataset N=47; CHI N=20, PHI N=27).
Arm/Group | CHI-patients | PHI-patients
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/27
Serious Adverse Events (participants affected / at risk) | 7/20 | 8/27
Other Adverse Events (participants affected / at risk) | 20/20 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHI-patients (N=20) | PHI-patients (N=27)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Cerebral infarction (Vascular disorders) | 0 (0) | 1 (1)
Basal ganglia stroke (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Renal stone removal (Surgical and medical procedures) | 0 (0) | 1 (2)
Hip arthroplasty (Surgical and medical procedures) | 2 (3) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Follow-up-report
Renal stone removal (Surgical and medical procedures) | 0 (0) | 1 (1) — Follow-up report (to reported Nephrolithiasis)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) — Hospitalization due to suspected urolithiasis (not confirmed)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHI-patients (N=20) | PHI-patients (N=27)
Nasopharyngitis (Infections and infestations) | 11 (26) | 14 (30)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Acute hepatitis C (Infections and infestations) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 0 (0) | 2 (2)
Anal chlamydia infection (Infections and infestations) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Bronchitis (Infections and infestations) | 4 (7) | 5 (6)
Chlamydial infection (Infections and infestations) | 0 (0) | 3 (3)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Depression (Psychiatric disorders) | 3 (4) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 10 (20)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Epididymitis (Infections and infestations) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (6) | 5 (6)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Folliculitis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (4)
Gastrointestinal viral infectio (Infections and infestations) | 2 (2) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 3 (3)
Gonorrhoea (Infections and infestations) | 0 (0) | 2 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 0 (0) | 4 (6)
Herpes virus infection (Infections and infestations) | 0 (0) | 2 (3)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (4)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Ocular icterus (Hepatobiliary disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (3) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Proctitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 4 (5) | 3 (4)
Sleep disorder (Psychiatric disorders) | 4 (4) | 3 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Syphilis (Infections and infestations) | 3 (9) | 8 (11)
Tonsillitis (Infections and infestations) | 2 (4) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 2 (2)
Urethritis gonococcal (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 (8) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT00908544/Prot_SAP_000.pdf